CLINICAL TRIAL: NCT05134480
Title: Diabetes Endothelial Keratoplasty Study (DEKS): Impact of Diabetes on Corneal Transplant Success and Endothelial Cell Loss
Brief Title: Impact of Donor Diabetes on DMEK Success and Endothelial Cell Loss
Acronym: DEKS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Collaborators: Jaeb Center for Health Research (Other); National Eye Institute (NEI) (NIH)
Responsible Party: Principal Investigator, Jonathan Lass, MD, Study Chair, Case Western Reserve University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DEKS; 1UG1EY030039-01A1 (NIH); 1UG1EY030030-01A1 (NIH)
Record Dates: First submitted 2021-11-13; First posted 2021-11-26 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Corneal Endothelial Decompensation; Fuchs' Endothelial Dystrophy
MeSH Terms: conditions — Fuchs' Endothelial Dystrophy

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, double-masked (participant and clinical site) clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The participants and the clinical site staff, including the investigators and outcomes assessor will be masked to all donor tissue parameters except storage solution.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cornea from donor with diabetes (Active Comparator): Participant will be assigned a cornea recovered from a donor with diabetes.
  Interventions: Procedure: Descemet membrane endothelial keratoplasty
- Cornea from donor without diabetes (Active Comparator): Participant will be assigned a cornea recovered from a donor without diabetes.
  Interventions: Procedure: Descemet membrane endothelial keratoplasty

INTERVENTIONS:
Procedure: Descemet membrane endothelial keratoplasty — cornea transplant procedure to replace dysfunctional endothelial cell layer

SUMMARY:
This double-masked multi-center trial will evaluate the association of diabetes in the cornea donor with transplant success and loss of endothelial cells through 1 year following Descemet membrane endothelial keratoplasty (DMEK). Study eyes are assigned to receive either a cornea from a donor without diabetes or a cornea from a donor with diabetes.

DETAILED DESCRIPTION:
This study will address concerns about the suitability of corneas from donors with diabetes for use with DMEK through a prospective, masked, multi-center clinical trial in which the donor corneas are assigned by diabetes status in the same distribution proportion (2:1 distribution of tissue from donors without diabetes to tissue from donors with diabetes) currently used in the USA. The DEKS will assess graft success and endothelial cell density through 1 year following DMEK to determine whether the surgical success rate with corneas from donors with well characterized diabetes (including post-mortem hemoglobin A1c (HbA1c) and advanced glycation end products (AGE) testing) is inferior to the rate with donors without diabetes. The investigators hypothesize that the majority of donor corneas from individuals with diabetes will be suitable, but that a portion of donors with a higher diabetes severity scale, and/or poorer control based on HbA1c will have a greater risk for graft failure and endothelial cell loss. This study will also examine collected skin biopsies to determine whether high levels of AGE biomarkers in donor skin tissue - which quantifies disease severity over many years (and possibly coupled with elevated HbA1c levels) - is associated with greater risk for graft failure and cell loss. This novel approach to characterization of donor tissue can provide a paradigm shift in the risk assessment of transplanted corneas from diabetic donors. The effect of recipient diabetes on keratoplasty success and cell loss will also be studied in a rigorous manner to determine the potential combined effect of donor and recipient diabetes status.

In summary, this study is designed to determine if non-diabetic donor corneas are superior to diabetic donor corneas in terms of both graft success and endothelial cell density outcomes, with an additional specific aim to determine whether donors with a higher diabetes severity scale, and/or poorer control based on HbA1c are driving the effect. This study will also determine whether a high AGE/A1c metric is also associated with the potential superiority finding and establish a novel composite score (severity score, HbA1c and AGE/A1c) based on these metrics that can be used to identify high versus low risk diabetic donors. This distinction may enable eye banks to potentially utilize the majority of donors with diabetes for EK surgery, while excluding the severely affected donors with diabetes.

ELIGIBILITY:
Participant Inclusion Criteria:

1. Age range 30- < 91 years with minimum life expectancy of at least 1 year
2. Willingness to return to study site for follow up at 1 month and 1 year
3. Fluent in English or Spanish
4. Willingness to have fingerstick blood sample collected to determine HbA1c level at entry and at 1 year. The participant must agree to have their primary care provider contacted (or an appropriate referral provided) if they were not known to have diabetes and the HbA1c suggests they may have diabetes. Similarly, if already known to have diabetes and the HbA1c is high, the participant must agree to have their primary care provider contacted or an appropriate referral provided.
5. Has at least one eye clinically recommended for DMEK that is able to be scheduled for DMEK between 5 to 90 days after enrollment. If second eye is enrolled, it must be scheduled for DMEK between 7 days and 6 months after DMEK on the first eye.
6. Has a condition related to endothelial dysfunction which will be treated by DMEK. Eligible indications for DMEK include:

   1. Presence of Fuchs endothelial corneal dystrophy (FECD) meeting at least one of the following: phakic FECD with or without cataract (triple procedure including DMEK for FECD, cataract extraction and posterior chamber intraocular lens implantation (IOL) is allowed)
   2. pseudophakic FECD with posterior capsule supported, sulcus supported, or scleral-fixated posterior chamber IOL
   3. pseudophakic corneal edema with posterior capsule supported, sulcus supported, or scleral-fixated posterior chamber IOL without FECD
   4. failed Descemet stripping automated endothelial keratoplasty (DSAEK) or DMEK originally performed for the same indications above without current exclusionary criteria, as described below

Exclusion Criteria:

1. Pregnant or planning to become pregnant prior to the DMEK study surgery, based on verbal report.
2. Lack cognitive capacity such that consent could not be provided.
3. Presence of a condition that has a high probability for failure (e.g., failed penetrating keratoplasty, uncontrolled uveitis)
4. Stromal vascularization that will impede assessment of recipient stroma clarity
5. Other primary endothelial dysfunction conditions including posterior polymorphous corneal dystrophy and congenital hereditary corneal dystrophy.
6. Indication for surgery that is not suitable for DMEK (e.g, keratoconus, stromal dystrophies and scars)
7. Aphakic corneal edema with or without FECD
8. Anterior chamber IOL in study eye prior to DMEK or planned placement of anterior chamber IOL during DMEK
9. Presence of vitreous in the anterior chamber
10. Planned IOL exchange of an anterior chamber IOL with a posterior chamber IOL in study eye at time of study DMEK
11. Pre-operative central sub-epithelial or stromal scarring that could impact post-operative recipient stromal clarity assessment
12. Presence of anterior synechiae
13. Peripheral anterior synechiae in the angle greater than a total of three clock hours
14. Uncontrolled glaucoma with or without prior filtering surgery, tube shunt placement, or MIGS. Uncontrolled glaucoma is defined as intraocular pressure > 25mm Hg.
15. Controlled glaucoma with prior tube shunt placement for glaucoma (controlled glaucoma with minimally invasive glaucoma surgery (MIGS) or trabeculectomy is allowed)
16. Fellow eye visual acuity < 20/200 due to an ocular condition other than a cornea disease that would be a candidate for DMEK
17. Intraocular pressure <8 mmHg
18. Topical Rho kinase inhibitor, including netarsudil, used within 1 month prior to study entry and anticipated during the course of the study
19. Fellow eye enrolled in the DEKS that has met study-criteria for graft failure.

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1097 (Actual)
Dates: Start 2022-01-21 (Actual); Primary Completion 2025-07-15 (Actual); Study Completion 2025-09-15 (Actual)

PRIMARY OUTCOMES:
Graft failure | 1 year
  Graft failure is defined as the occurrence of one of the following: a graft which requires replacement for any reason or the recipient cornea remains cloudy after surgery without clearing for 8 weeks or longer

SECONDARY OUTCOMES:
Endothelial cell density | 1 year
  Central corneal endothelial cell density assessed with specular microscopy

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Lass, MD, Study Chair — Case Western Reserve University
Locations (2):
- United States (2):
  - Price Vision Group, Indianapolis, Indiana
  - Verdier Eye Center, Grand Rapids, Michigan

IPD SHARING:
Plan to Share IPD: Yes
Data collected for this study will be analyzed and stored at the Jaeb Center for Health Research. After the study is completed, the de-identified, archived data will be made publicly available. Further, some data and images may be requested and shared with other researchers under a Data Use Agreement as a limited data set, since other than date of collection, there are no other identifiable elements. No additional identifying information shall be provided in a manner that would make the human subjects readily identifiable.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be made available indefinitely after publication of the study results, which is anticipated by July, 2030.

REFERENCES:
- [Derived] Lass JH, Benetz BA, Verdier DD, Szczotka-Flynn LB, Bauza CE, Reed ZW, Greiner MA, Mian SI, Patel SV, Pramanik S, Price FW Jr, Soper MC, Terry MA, Titus MS, Kollman C, Beck RW, Price MO; Diabetes Endothelial Keratoplasty Study Group. Endothelial Cell Loss 1 Year After Successful DMEK in the Diabetes Endothelial Keratoplasty Study: A Randomized Clinical Trial. JAMA Ophthalmol. 2025 Dec 1;143(12):1053-1060. doi: 10.1001/jamaophthalmol.2025.4261. PMID 41105099
- [Derived] Price FW Jr, Szczotka-Flynn LB, Price MO, Bauza CE, Reed ZW, Arafah BM, Greiner MA, Johnson PJ, Keeler DB, Mian SI, Patel SV, Pramanik S, Soper MC, Terry MA, Titus MS, Verdier DD, Kollman C, Beck RW, Lass JH; Diabetes Endothelial Keratoplasty Study Group. Donor Diabetes and 1-Year Descemet Membrane Endothelial Keratoplasty Success Rate: A Randomized Clinical Trial. JAMA Ophthalmol. 2025 Dec 1;143(12):1043-1051. doi: 10.1001/jamaophthalmol.2025.4253. PMID 41105094
- [Derived] Price MO, Szczotka-Flynn LB, Bauza CE, Reed ZW, Benetz BA, Greiner MA, Verdier DD, Soper MC, Titus MS, Monnier VM, Arafah BM, Kollman C, Beck RW, Lass JH; Writing Committee for the Diabetes Endothelial Keratoplasty Study Group. Diabetes Endothelial Keratoplasty Study: Methods and Impact on the Use of Corneas From Donors With Diabetes for Descemet Membrane Endothelial Keratoplasty. Cornea. 2026 Mar 1;45(3):312-321. doi: 10.1097/ICO.0000000000003776. Epub 2025 Jan 9. PMID 39808526

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-01-26): https://cdn.clinicaltrials.gov/large-docs/80/NCT05134480/Prot_SAP_002.pdf
  • Informed Consent Form (2023-02-06): https://cdn.clinicaltrials.gov/large-docs/80/NCT05134480/ICF_001.pdf